CLINICAL TRIAL: NCT05963542
Title: SoundMind Trial: a Randomized Controlled Trial of Online Acceptance and Commitment Therapy and Sound Therapy for Tinnitus
Brief Title: Efficacy of Online Acceptance and Commitment Therapy and Sound Therapy for Patients With Tinnitus and Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023066-1
Record Dates: First submitted 2023-07-16; First posted 2023-07-27 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Tinnitus; Insomnia
MeSH Terms: conditions — Tinnitus; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT + sound therapy group (Experimental): The combined treatment group will receive Internet-delivered guided self-help tinnitus treatment based on ACT combined with customized sound therapy.
  The online ACT program includes 8 modules of structured self-help material over 8 weeks. Each module includes information, exercises, and homework. The self-help material covers the six core processes of ACT: acceptance, cognitive defusion, being present, self-as-context, values, and committed action, emphasizing psychological flexibility.
  Customized sound therapy will be provided by the Fudan Tinnitus Relieving System (FTRS) app. Participants will listen to tailor-made music through the app for more than two hours per day.
  Interventions: Behavioral: ACT for tinnitus; Other: Customized sound therapy
- sound therapy group (Active Comparator): The single treatment group will receive customized sound therapy provided by the FTRS app for more than two hours per day.
  Interventions: Other: Customized sound therapy

INTERVENTIONS:
Behavioral: ACT for tinnitus — The intervention will be based on the ACT model and adjusted for tinnitus.
  Arms: ACT + sound therapy group
Other: Customized sound therapy — The music will be modulated through a smartphone app using a set program to generate customized tinnitus relieving sound.

SUMMARY:
Considering the lack of evidence on the effects of combining acceptance and commitment therapy (ACT) with customized sound therapy for tinnitus-related insomnia patients, investigators designed this single-blind, 6-months randomized, controlled trial with two parallel groups. One is the ACT + sound therapy group, and the other is the sound therapy group.

DETAILED DESCRIPTION:
Insomnia is one of the most frequent and severe comorbidities in patients with tinnitus and is highly relevant for the perceived tinnitus severity. Both tinnitus and insomnia significantly affect the quality of life of patients and represent a huge burden to society. While interventions exist to alleviate tinnitus distress, they often do not address sleep disturbances in tinnitus patients. Patients affected by tinnitus and insomnia suffer from long-term functional and psychological problems. Sound therapy is widely used to treat tinnitus, often combined with education and counseling, and can effectively improve the quality of life. In addition, acceptance and commitment therapy (ACT) for tinnitus improves both tinnitus and sleep. However, there is a lack of evidence on the effects of combining ACT with sound therapy for tinnitus-related insomnia patients.

To fully characterize tinnitus patients, standardized measures of tinnitus and insomnia are essential. These measures include pure tone audiometry (PTA), acoustic immittance (AI), tinnitus pitch matching (PM) and loudness matching (LM), minimum masking level (MML), tinnitus handicap inventory (THI), insomnia severity index (ISI), and hospital anxiety and depression scale (HADS).

Investigators hypothesize that the combination of ACT and sound therapy will be superiority to sound therapy alone in reducing tinnitus distress.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18 and 80 years old.
2. Experiencing subjective tinnitus for at least 3 months.
3. A score of 38 or more on THI.
4. A score of 15 or more on ISI.
5. 55 dB HL or less on the average pure tone threshold (0.5, 1, 2kHz) of the worse ear.
6. Ability to read and write in Chinese and use a smartphone with an internet connection to work with text material.

Exclusion Criteria:

1. Pulsatile tinnitus and objective tinnitus.
2. Organic sleep disorders.
3. Other diseases that need to be treated first (e.g., infections, tumors, otosclerosis, Meniere's disease, the acute stage of sudden sensorineural hearing loss).
4. Severe mental illness.
5. Undergoing other research that may affect tinnitus and sleep.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | 2 months from baseline
  The THI questionnaire, widely used in research, including functional, emotional, and catastrophic subscales. It consists of 25 questions, and answers are rated on a "yes" (4 points), "sometimes" (2 points), and "no" (0 points) scale. The total score is calculated by adding up the scores for all questions and classifying the severity of tinnitus as no handicap (0-16), mild handicap (18-36), moderate handicap (38-56), and severe handicap (58-100).
Tinnitus Handicap Inventory (THI) | 3 months from baseline
  The THI questionnaire, widely used in research, including functional, emotional, and catastrophic subscales. It consists of 25 questions, and answers are rated on a "yes" (4 points), "sometimes" (2 points), and "no" (0 points) scale. The total score is calculated by adding up the scores for all questions and classifying the severity of tinnitus as no handicap (0-16), mild handicap (18-36), moderate handicap (38-56), and severe handicap (58-100).
Tinnitus Handicap Inventory (THI) | 6 months from baseline
  The THI questionnaire, widely used in research, including functional, emotional, and catastrophic subscales. It consists of 25 questions, and answers are rated on a "yes" (4 points), "sometimes" (2 points), and "no" (0 points) scale. The total score is calculated by adding up the scores for all questions and classifying the severity of tinnitus as no handicap (0-16), mild handicap (18-36), moderate handicap (38-56), and severe handicap (58-100).

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | 2 months from baseline
  ISI is a self-report questionnaire that assesses the severity and impact of insomnia over the last two weeks. The questionnaire consists of seven items that evaluate the severity of sleep onset, sleep maintenance, early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by sleep difficulties. Each item is scored on a 0-4 scale, and the total score is interpreted as the absence of insomnia (0-7), sub-threshold insomnia (8-14), moderate insomnia (15-21), and severe insomnia (22-28).
Insomnia Severity Index (ISI) | 3 months from baseline
  ISI is a self-report questionnaire that assesses the severity and impact of insomnia over the last two weeks. The questionnaire consists of seven items that evaluate the severity of sleep onset, sleep maintenance, early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by sleep difficulties. Each item is scored on a 0-4 scale, and the total score is interpreted as the absence of insomnia (0-7), sub-threshold insomnia (8-14), moderate insomnia (15-21), and severe insomnia (22-28).
Insomnia Severity Index (ISI) | 6 months from baseline
  ISI is a self-report questionnaire that assesses the severity and impact of insomnia over the last two weeks. The questionnaire consists of seven items that evaluate the severity of sleep onset, sleep maintenance, early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by sleep difficulties. Each item is scored on a 0-4 scale, and the total score is interpreted as the absence of insomnia (0-7), sub-threshold insomnia (8-14), moderate insomnia (15-21), and severe insomnia (22-28).
Sleep Onset Latency (SOL) | 2 months from baseline
  SOL will be estimated with actigraphy. Actigraphy is a small watch worn on the participant's non-dominant wrist that collects objective sleep parameters. Lower score indicates better sleep.
Sleep Onset Latency (SOL) | 3 months from baseline
  SOL will be estimated with actigraphy. Actigraphy is a small watch worn on the participant's non-dominant wrist that collects objective sleep parameters. Lower score indicates better sleep.
Sleep Onset Latency (SOL) | 6 months from baseline
  SOL will be estimated with actigraphy. Actigraphy is a small watch worn on the participant's non-dominant wrist that collects objective sleep parameters. Lower score indicates better sleep.
Wake After Sleep Onset (WASO) | 2 months from baseline
  WASO will be estimated with actigraphy. Actigraphy is a small watch worn on the participant's non-dominant wrist that collects objective sleep parameters. Lower score indicates better sleep.
Wake After Sleep Onset (WASO) | 3 months from baseline
  WASO will be estimated with actigraphy. Actigraphy is a small watch worn on the participant's non-dominant wrist that collects objective sleep parameters. Lower score indicates better sleep.
Wake After Sleep Onset (WASO) | 6 months from baseline
  WASO will be estimated with actigraphy. Actigraphy is a small watch worn on the participant's non-dominant wrist that collects objective sleep parameters. Lower score indicates better sleep.
Sleep Efficiency (SE) | 2 months from baseline
  SE will be estimated with actigraphy. Actigraphy is a small watch worn on the participant's non-dominant wrist that collects objective sleep parameters. Higher score indicates better sleep.
Sleep Efficiency (SE) | 3 months from baseline
  SE will be estimated with actigraphy. Actigraphy is a small watch worn on the participant's non-dominant wrist that collects objective sleep parameters. Higher score indicates better sleep.
Sleep Efficiency (SE) | 6 months from baseline
  SE will be estimated with actigraphy. Actigraphy is a small watch worn on the participant's non-dominant wrist that collects objective sleep parameters. Higher score indicates better sleep.
Visual Analogue Scale (VAS) | 2 months from baseline
  Subjective perception of tinnitus loudness will be assessed using the VAS. Participants will be asked to rate the loudness of the tinnitus on a scale ranging from 0 (no tinnitus) to 10 (tinnitus could not be louder).
Visual Analogue Scale (VAS) | 3 months from baseline
  Subjective perception of tinnitus loudness will be assessed using the VAS. Participants will be asked to rate the loudness of the tinnitus on a scale ranging from 0 (no tinnitus) to 10 (tinnitus could not be louder).
Visual Analogue Scale (VAS) | 6 months from baseline
  Subjective perception of tinnitus loudness will be assessed using the VAS. Participants will be asked to rate the loudness of the tinnitus on a scale ranging from 0 (no tinnitus) to 10 (tinnitus could not be louder).
Hospital Anxiety and Distress Scale (HADS) | 2 months from baseline
  HADS is a 14-item self-report questionnaire with two 7-item subscales to assess symptoms of anxiety (HADS-A) and depression (HADS-D)[31]. Each item is scored from 0-3, with each subscale ranging from 0-21. A threshold value of 8 or greater for the HADS-A or HADS-D indicates clinically significant symptoms of anxiety or depression.
Hospital Anxiety and Distress Scale (HADS) | 3 months from baseline
  HADS is a 14-item self-report questionnaire with two 7-item subscales to assess symptoms of anxiety (HADS-A) and depression (HADS-D)[31]. Each item is scored from 0-3, with each subscale ranging from 0-21. A threshold value of 8 or greater for the HADS-A or HADS-D indicates clinically significant symptoms of anxiety or depression.
Hospital Anxiety and Distress Scale (HADS) | 6 months from baseline
  HADS is a 14-item self-report questionnaire with two 7-item subscales to assess symptoms of anxiety (HADS-A) and depression (HADS-D)[31]. Each item is scored from 0-3, with each subscale ranging from 0-21. A threshold value of 8 or greater for the HADS-A or HADS-D indicates clinically significant symptoms of anxiety or depression.
Tinnitus Acceptance Questionnaire (TAQ) | 2 months from baseline
  TAQ consists of 12 items divided into two factors: activity engagement and tinnitus suppression, and is widely used as a measure of experiential avoidance/acceptance in relation to tinnitus. The total score is 72, with higher scores indicating a higher level of tinnitus-related acceptance.
Tinnitus Acceptance Questionnaire (TAQ) | 3 months from baseline
  TAQ consists of 12 items divided into two factors: activity engagement and tinnitus suppression, and is widely used as a measure of experiential avoidance/acceptance in relation to tinnitus. The total score is 72, with higher scores indicating a higher level of tinnitus-related acceptance.
Tinnitus Acceptance Questionnaire (TAQ) | 6 months from baseline
  TAQ consists of 12 items divided into two factors: activity engagement and tinnitus suppression, and is widely used as a measure of experiential avoidance/acceptance in relation to tinnitus. The total score is 72, with higher scores indicating a higher level of tinnitus-related acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Huawei Li, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Fudan University Eye Ear Nose and Throat Hospital, Otorhinolaryngology Department, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang X, Tang D, Sun S, Li H. SoundMind Trial: a study protocol for a randomised controlled trial for online acceptance and commitment therapy and sound therapy for tinnitus. BMJ Open. 2024 Oct 17;14(10):e080863. doi: 10.1136/bmjopen-2023-080863. PMID 39419615